CLINICAL TRIAL: NCT06588738
Title: A Multicenter, Randomized, Double-Blind, Placebo and Active Comparator Controlled Phase 3 Study in Patients With Moderate to Severe Plaque Psoriasis to Evaluate the Efficacy and Safety of ESK-001 (ONWARD2)
Brief Title: A Study in Patients With Moderate to Severe Plaque Psoriasis to Evaluate the Efficacy and Safety of ESK-001
Acronym: ONWARD2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESK-001-017
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ESK-001 (Experimental): ESK-001 administered as an oral tablet
  Interventions: Drug: ESK-001
- Placebo (Placebo Comparator): Matching oral placebo
  Interventions: Drug: Placebo
- Apremilast (Active Comparator): Apremilast administered as an oral capsule
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: ESK-001 — ESK-001
  Arms: ESK-001
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Apremilast — Apremilast
  Arms: Apremilast

SUMMARY:
The goal of this clinical trial is to learn if ESK-001 works to treat moderate to severe plaque psoriasis. The main questions it aims to answer are:

* Does ESK-001 reduce the severity of people's psoriasis?
* How safe is ESK-001 in people with moderate to severe plaque psoriasis?

The study includes 2 comparators: a placebo control (a 'dummy' tablet that does not contain the medicine ESK-001 but looks just like it) and an active control (apremilast, which is a medicine approved to treat psoriasis).

People taking part in this study must be men or women aged at least 18 years and have had plaque psoriasis for at least 6 months, currently moderate to severe.

Participants will:

* take drug every day for 24 weeks.
* visit the clinic for checkups and tests.
* fill out questionnaires about their psoriasis, itch severity, and change in quality of life.
* be assessed for health issues and side effects, physical examinations, vital signs, heart electrical activity measurements, and psychological health.
* provide blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age ≥18 years
2. Diagnosis of plaque psoriasis for ≥6 months
3. Plaques covering ≥10% of BSA
4. PASI ≥12
5. sPGA ≥3
6. Women of childbearing potential (WOCBP) and males who are sexually active with WOCBP must agree to adhere to highly effective methods of contraception

Exclusion Criteria:

1. Nonplaque psoriasis or other inflammatory skin conditions
2. Immune-mediated conditions commonly associated with psoriasis (eg inflammatory bowel disease). Patients with psoriatic arthritis may participate
3. Pregnant, lactating, or planning to get pregnant during the study
4. Use of drugs prior to Study Day 1 that treat or may affect psoriasis:

   * Topical within 2 weeks
   * Phototherapy or any systemic treatments within 4 weeks
   * Any biologic agent targeted to IL-12 or IL-23 within 6 months, oral IL-12 or IL-23 or TNFα inhibitor within 2 months, or IL-17 within 4 months
   * Systemic immunosuppressants or immunomodulatory drugs within 4 weeks
   * Modulators of B cells within 6 months, or T cells within 3 months
   * JAK inhibitors or TYK2 inhibitors within 4 weeks
   * PDE4 inhibitor within 2 months
   * Any investigational agent, within 30 days or 5 half-lives or is currently enrolled in an investigational study
5. Lack of clinical response to a TYK2, IL-12, or IL-23 targeted psoriasis treatment
6. Patients with QTcF >450 msec (males) or >470 msec (females) at Screening
7. Unstable cardiovascular disease, defined as a recent clinical deterioration or a cardiac hospitalization within the last 3 months
8. Evidence of recent or recurrent herpes zoster or herpes simplex viral infection
9. Evidence of active infection or positive test result for hepatitis B, hepatitis C, HIV or TB
10. History of serious bacterial, fungal, or viral infections that led to hospitalization, or any recent serious infection requiring antibiotic treatment
11. Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the patient's immune status
12. Lab abnormalities indicating significant renal, hepatic or bone marrow dysfunction
13. History of any immune-mediated or inflammatory medical condition for which patient requires current systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether ESK-001 reduces the severity of psoriasis by 75% (using the PASI) or by at least 2 points (using sPGA score) compared to placebo | 16 weeks
  Proportion of patients achieving ≥75% reduction in PASI score. Proportion of patients achieving a score of 0 or 1 on sPGA.

SECONDARY OUTCOMES:
To compare the Psoriasis Area and Severity Index (PASI-90 and PASI-100) between ESK-001 and placebo or apremilast | 24 weeks
  Proportion of patients achieving of ≥90% or 100% reduction in PASI
To compare the Psoriasis Area and Severity Index (PASI-75) between ESK-001 and apremilast | 24 weeks
  Proportion of patients achieving of ≥75% reduction in PASI
To compare the Static Physician's Global Assessment (sPGA-0/1) between ESK-001 and apremilast | 24 weeks
  Proportion of patients achieving a score of 0 or 1 on sPGA
To compare the affected body surface area (%BSA) between ESK-001 and placebo or apremilast | 24 weeks
  Change from baseline in %BSA
To compare the scalp specific Physician's Global Assessment (ssPGA) between ESK-001 and placebo or apremilast | 24 weeks
  Proportion of patients achieving a score of 0 or 1 on ssPGA
To compare the Psoriasis Symptoms and Signs Diary (PSSD) between ESK-001 and placebo or apremilast | 24 weeks
  Proportion of patients achieving a score of 0
To compare the Dermatology Life Quality Index (DLQI) between ESK-001 and placebo or apremilast | 24 weeks
  Proportion of patients achieving a score of 0 or 1
To compare the Pruritus numeric rating scale (NRS) between ESK-001 and placebo | 24 weeks
  Change from baseline in Pruritus NRS (scale is from 0 (no pain) to 10 (severe pain)).
Proportion of patients with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 24 weeks
  Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)
To characterize the pharmacokinetics of ESK-001 | 24 weeks
  Maximum [Cmax] and minimum [Cmin] plasma concentration

CONTACTS AND LOCATIONS:
Locations (125):
- United States (43):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Zenith Research Inc., Beverly Hills, California
  - Raoof MD, Encino, California
  - Long Beach Research Institute, Long Beach, California
  - Dermatology Research Associates, Los Angeles, California
  - Empire Clinical Research - Pomona, Pomona, California
  - Integrative Skin Science and Research, Sacramento, California
  - UC San Diego, San Diego, California
  - Southern California Clinical Research, Santa Ana, California
  - Clinical Science Institute Dermatology Institute, Santa Monica, California
  - FXM Clinical Research Ft. Lauderdale LLC, Fort Lauderdale, Florida
  - Direct Helpers Research Center (DHRC), Hialeah, Florida
  - AppleMed Research Group under WCG, Miami, Florida
  - FAX Pharma Clinical Research Inc, Miami, Florida
  - FXM Clinical Research - Miami LLC, Miami, Florida
  - Las Mercedes Medical Research, Miami, Florida
  - FXM Clinical Research Miramar LLC, Miramar, Florida
  - Renstar Medical Research, Ocala, Florida
  - DS Research of Southern Indiana, Clarksville, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - DS Research of Kentucky, Louisville, Kentucky
  - Michigan Center for Research Company, Clarkston, Michigan
  - Henry Ford Medical Center - Farmington Road, Detroit, Michigan
  - Revival Research Institute, Troy, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Associated Skin Care Specialists - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Schlessinger MD, Omaha, Nebraska
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - NYC Health and Hospitals Elmhurst, Elmhurst, New York
  - Pioneer Clinical Research NY, New York, New York
  - Cameron Dermatology, New York, New York
  - DermResearchCenter of New York, Stony Brook, New York
  - Asheville Clinical Trials, Asheville, North Carolina
  - WDC Cosmetic and Research, Wilmington, North Carolina
  - Optima Research Boardman, Boardman, Ohio
  - Clinical Partners LLC, Johnston, Rhode Island
  - Modern Research Associates PLLC, Dallas, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Progressive Clinical Research - San Antonio, San Antonio, Texas
  - Center for Clinical Studies (CCS) - Webster/Clear Lake Location, Webster, Texas
  - Jordan Valley Dermatology, South Jordan, Utah
- Klinik Hietzing, Vienna, Vienna, Austria
- Canada (17):
  - Beacon Dermatology, Calgary, Alberta
  - Alberta DermaSurgery, Edmonton, Alberta
  - VIDA Dermatology/VIDA Clinical Research, Edmonton, Alberta
  - CaRe Clinic Red Deer, Red Deer, Alberta
  - Skincare Studio, St. John's, Newfoundland and Labrador
  - CCA Medical Research Corp, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - SKiN Health, Cobourg, Ontario
  - Guelph Dermatology Research, Guelph, Ontario
  - Mediprobe Research, London, Ontario
  - Clear Skin Dermatology, Newmarket, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Rejuvination Dermatology Oakville, Oakville, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Innovaderm, Montreal, Quebec
  - SkinSense Medical Research, Saskatoon, Saskatchewan
- Estonia (4):
  - Innomedica, Tallinn, Harju
  - Tartu University Hospital, Tartu, Tartu
  - Center for Clinical and Basic Research AS, Tallinn
  - Kliiniliste Uuringute Keskus OU, Tartu
- France (3):
  - CHU de Rouen, Rouen, Normandy
  - Centre Azur Nice, Nice
  - Polyclinique de Courlancy, Reims
- Germany (13):
  - Universitatsklinikum Erlangen, Erlangen, Bavaria
  - Rosenpark Research, Darmstadt, Hesse
  - Klinikum Oldenburg, Oldenburg, Lower Saxony
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Hautarztpraxis Dr Niesmann and Dr Othlinghaus, Bochum, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Dermatologische Praxis Dres Quist, Mainz, Rhinelkand-Palatinate
  - Praxis fur Dermatologie und Venerologie, Dresden, Saxony
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - ISA - Interdisciplinary Study Association GmbH, Berlin, State of Berlin
  - MVZ DermaKiel GmbH, Kiel
  - Haut Ambulatorium Magdeburg, Magdeburg
  - KliFOs Klinische Forschung Osnabruck, Osnabrück
- Hungary (8):
  - Bacs Kiskun County Teaching Hospital, Kecskemét, Bács-Kiskun county
  - Borgyogyaszati Klinika Debreceni Egyetem Orvos es Egeszsegtudomenyi Centrum, Debrecen, Hajdú-Bihar
  - DERMA B Kft, Debrecen, Hajdú-Bihar Megye
  - DermaMed Research Kf, Békés, Oroshaza
  - Uno Medical Trials Kft, Budapest
  - Orvostudomanyi Kutato es Fejleszto Kft, Debrecen
  - Allergo Derm Bakos Kft, Szolnok
  - Medmare Bt, Veszprém
- Sheba Tel HaShomer Medical Centre, Ramat Gan, Israel
- Latvia (7):
  - Semigallia Ltd, Kuldīga, Kuldigas
  - Smite Aija Medical Practice in Dermatology Venereology, Talsi, Talsi
  - Riga 1st Hospital, Riga
  - Med Art Clinic, Riga
  - Veselibas Centrs 4, Riga
  - SIA Veseliba un estetika, Riga
  - Veselibas Centrs 4 Filiale Dermatologijas Klinika, Riga
- Poland (18):
  - FutureMeds Krakow, Krakow, Lesser Poland Voivodeship
  - Luxderm, Lublin, Lublin Voivodeship
  - Centrum Medyczne dr Rajzer Spolka Zoo, Krakow, Malopolska
  - RCMed Oddział Sochaczew, Sochaczew, Masovian Voivodeship
  - Clinical Best Solutions, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship
  - Klinika Dermatologii Uniwersytecki Szpital Kliniczny im F Chopina, Rzeszów, Podkarpackie Voivodeship
  - Specderm, Bialystok, Podlaskie Voivodeship
  - Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - Pratia Katowice, Katowice, Silesian Voivodeship
  - Research Solutions, Katowice, Silesian Voivodeship
  - Care Clinic Katowice, Katowice
  - Zanamed Medical Clinic Sp z o o, Lublin
  - MTZ Clinical Research Sp z o o, Warsaw
  - Klinika Ambroziak Dermatologia Kliniczna, Warsaw
  - dermMedica, Wroclaw
  - Dermoklinika, Lodz, Łódź Voivodeship
  - FutureMeds Lodz, Lodz, Łódź Voivodeship
- Puerto Rico (4):
  - GCM Medical Group PSC Hato Rey Site, San Juan, PR
  - Centro Reumatologico de Caguas, Caguas, Puerto Rico
  - Ponce Medical School Foundation Inc, Ponce, Puerto Rico
  - Clinical Research Puerto Rico, Ponce, Puerto Rico
- Spain (6):
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - University General Hospital Dr Balmis, Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital de Manises, Manises
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor Alumis Inc. is a clinical-stage biopharmaceutical company that has not yet adopted an Individual Participant Data (IPD) sharing plan.